CLINICAL TRIAL: NCT04569019
Title: Attitudes Towards Influenza Vaccinations Among the Healthcare Workers of the University Clinical Center of the Medical University of Warsaw
Brief Title: Attitudes Towards Influenza Vaccinations Among the Healthcare Workers of Medical University of Warsaw
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Dominika Rykowska, MD, Medical University of Warsaw
Other Study IDs: AKBE/118/2020
Record Dates: First submitted 2020-09-23; First posted 2020-09-29 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Vaccnation in HCW
Keywords: Medicine Vaccinations among healthcare professionals ,Vaccinations against influenza ,COVID19 pandemic and its impact on influenza vaccination coverage

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Health care workers: The study will be conducted among UCKWUM healthcare professionals, i.e. doctors, nurses, paramedics, laboratory workers, pharmacists, and administration workers. Based on previous research, the group should include at least 200 participants
  Interventions: Other: Vacciantion status in health care workers

INTERVENTIONS:
Other: Vacciantion status in health care workers — Education among HCW about benefits of influenza vaccination. Using posters, email, conversations, informations about vaccination used during vaccination Vaccinating during working hours Vaccinating for free Vaccinating inside departments ( not in special clinic)

SUMMARY:
The study will be conducted in the UCKWUM teaching hospital in Warsaw between 2020 and 2022. The study group will be comprised of UCKWUM healthcare professionals All employees willing to participate in the study will receive an anonymous questionnaire on attitudes towards influenza vaccination . We will distribute information posters of the National Programme for Combating Influenza as part of the educational programme. In order to increase the effectiveness of the educational campaign, we will also send information e-mails, using the internal hospital e-mail system and conduct a series of online training courses to present the latest international reports on influenza vaccinations among health care professionals [CITATION Abr10 \l 1045].

Considering the fact that lack of time [CITATION Kus11 \l 1045] is the most common reason for not getting vaccinated against influenza among healthcare professionals, we will provide this group with an opportunity to receive free influenza vaccination during working hours at the UCKWUM hospital. Information about the possibility of vaccination will be provided in the form of e-mails (mailings) to hospital employees (internal hospital e-mail system), letters of information submitted to the offices of individual departments, and information posters.

The effectiveness of the educational programme will be assessed by re-administering the anonymous questionnaires after the influenza season, also by means of internal hospital e-mail system.

ELIGIBILITY:
Inclusion Criteria:

* Health Care worker of UCK WUM in Warsaw

Exclusion Criteria:

* non

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study will be conducted among UCKWUM healthcare professionals, i.e. doctors, nurses, paramedics, laboratory workers, pharmacists, and administration workers. Based on previous research, the group should include at least 200 participants
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-08-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Assesment of vaccination indeks in the hsopital by using questionare | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Warsaw Medical Uniwerity, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rykowska D, Sobierajski T, Okarska-Napierala M, Wanke-Rytt M, Kuchar E. Influenza vaccination from the perspective of health care workers at university hospitals. PLoS One. 2023 Jul 21;18(7):e0288470. doi: 10.1371/journal.pone.0288470. eCollection 2023. PMID 37478110